CLINICAL TRIAL: NCT01830023
Title: Vitality Trial - Sampling Examination Data
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-28
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cardiac Event
Keywords: cardiac ultrasound; vitality; data; patients; examined
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac ultrasound examination
  Interventions: Device: cardiac ultrasound examination

INTERVENTIONS:
Device: cardiac ultrasound examination — cardiac ultrasound examination to examine the vitality

SUMMARY:
This study´s aim is to collect data of vitality diagnosis. A cardiac ultrasound examination will be done and the data will be compared to the other examinations.

ELIGIBILITY:
Inclusion Criteria:

* MRI exmination outcome: positive Late Enhancement, proof of infarction scars by contrast agent.

Exclusion Criteria:

* no exclusion criteria as patients are asked to participate after evaluating the MRI examination outcome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are examined in the department of cardiology, university hospital Aachen
Sampling Method: Non-Probability Sample
Enrollment: 2019 (Actual)
Dates: Start 2009-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
vitality data | 1 day (at time of examination)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, university hospital, Aacehn, North Rhine Westfalia, Germany